CLINICAL TRIAL: NCT01197651
Title: Aortenstent-Register Thorakale Aorta
Brief Title: Aortic-Stent-Register
Status: Completed | Type: Observational
Sponsor: Stiftung Institut fuer Herzinfarktforschung (Other)
Responsible Party: Sponsor
Other Study IDs: Aortenstent
Record Dates: First submitted 2010-09-07; First posted 2010-09-09 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Aortic Dissection
Keywords: Aorta; Aorta-Stent-Graft; Surgical operation; Aortic dissection
MeSH Terms: conditions — Aortic Dissection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aims of the aorta-stent-Registry are:

• participating hospitals (with audit) document all consecutive patients diagnosed with a disease of the distal thoracal aorta that receive one of the following therapies:

DETAILED DESCRIPTION:
1. Endovascular Aorta-Stent-Graft
2. Surgical operation of the distal thoracal aorta

   * Documentation of the indications, the procedural results and the clinical short- and long-term results of the endovascular and chirurgical treatment in day to day hospital routine.
   * Documentation of the operational risk (Euroscore)
   * Documentation of the technical enforcement of the procedure as well as the result of the intervention
   * Documentation of the hospital lethality and the non-fatal serious complications (Spinal Cord Ischemia, SCI, Stroke, TIA, high blood loss etc.)
   * Documentation of medication at hospital discharge
   * Documentation of long-term lethality and non-fatal serious complications (SCI, Stroke, TIA, major bleeding etc.) as well as hospitalization, re-intervention rates and medicinal drug therapy after 30 days, 1, 3 & 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with significant illness of the distal thoracal aorta (distal Aortic-dissection; TAA; penetrated ulcer; covered perforation; traumatically transection of the distal thoracal aorta) including those that receive an endovascular stent or an open surgical operation.

Exclusion Criteria:

* Missing signed informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients being treated in one of the participating hospitals because of a disease of the distal thoracal aorta
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2008-10; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
◦Documentation of the indications, the procedural results and the clinical short- and long-term results of the endovascular and chirurgical treatment in day to day hospital routine | Hospital-stay

CONTACTS AND LOCATIONS:
Overall Officials: Raimund Erbel, MD, Study Chair — Westdeutsches Herzzentrum Essen; Holger Eggebrecht, MD, Study Chair — Westdeutsches Herzzentrum Essen; Thomas Helmberger, MD, Study Chair — Klinikum Bogenhausen; Christoph Nienaber, MD, Study Chair — Universitätsklinikum Rostock; Hüseyin Ince, MD, Study Chair — Universitätsklinikum Rostock; Harald Mudra, MD, Study Chair — Klinikum Neuperlach; Ralf Zahn, MD, Study Chair — Klinikum Ludwigshafen; Jochen Senges, MD, Study Chair — Institut für Herzinfarktforschung Ludwigshafen an der Universität Heidelberg
Locations (8):
- Germany (8):
  - Herz-Zentrum Bad Krozingen, Bad Krozingen
  - Kerckhoff-Klinik GmbH, Bad Nauheim
  - Segeberger Kliniken GmbH, Bad Segeberg
  - Westdeutsches Herzzentrum Essen, Uniklinikum, Essen
  - Klinikum Ludwigshafen, Ludwigshafen
  - Universitätsklinikum Magdeburg, Magdeburg
  - Städt. Klinikum München GmbH, München
  - Universitätsklinikum Rostock, Rostock

IPD SHARING:
Plan to Share IPD: No